CLINICAL TRIAL: NCT04831827
Title: Promoting Equity Through Multicomponent Strategies for Cancer Screening and Follow-up (PREMiS)
Brief Title: Promoting Equity for Cancer Screening and Follow-up
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient study resources and change in practice.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Chyke A. Doubeni, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20-012010
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Colorectal (Colon or Rectal) Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigators will be blinded to study arm; research coordinators will not be blinded because it is not practical to do so, but steps will be taken to minimize their awareness about study hypotheses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IVR Reminder (Experimental): Participants will receive an interactive voice reminder
  Interventions: Other: IVR Reminder
- Personalized Phone Call Reminder (Active Comparator): Participants will receive a personalized phone call
  Interventions: Other: Phone call from research team
- Portal Message Only (Active Comparator): Participants will receive a online patient portal message reminder
  Interventions: Other: EHR Portal message

INTERVENTIONS:
Other: IVR Reminder — Participants will receive an interactive voice reminder (IVR) to complete mt-sDNA screening at day 7 and 21.
  Arms: IVR Reminder
Other: Phone call from research team — Patients will receive a scripted phone call from the research team to remind them to complete the mt-sDNA screening at day 7 and 21.
  Arms: Personalized Phone Call Reminder
Other: EHR Portal message — Patients will receive an EHR patient portal message with a scripted message to remind them to complete the mt-sDNA screening at day 7 and 21.
  Arms: Portal Message Only

SUMMARY:
This is a randomized trial to assess the efficacy of reminder mechanisms on colorectal cancer (CRC) screening uptake among a cohort of patients who were previously mailed a multitarget stool DNA (mt-sDNA) test and did not complete the screening. Patients will be identified as being due for CRC screening and will be mailed a mt-sDNA kit to their home. Patients who do not complete screening with mt-sDNA within 30 days will be identified and randomized into one of three study arms to receive reminders to complete the mt-sDNA screening. The primary outcome is the rate of completion of screening for colorectal cancer with mt-sDNA test.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third leading cause of cancer-related death in the United States, and screening has been shown to reduce mortality from CRC. Screening is underutilized in the United States, particularly in some communities such as Blacks/African Americans, American Indians/Alaskan Natives, and rural populations, contributing to disparities in mortality.

For CRC screening, mt-sDNA testing is one of several tests that are recommended by the United States Preventive Services Task Force (USPSTF). As part of a quality improvement program at our institution, those who are due for CRC screening are identified using a validated electronic algorithm and a kit is mailed directly to each patient. Our intervention is initiated on non-respondents to the mailed mt-sDNA outreach by testing the use of a technology-enabled reminder system.

Thirty days after being mailed a mt-sDNA kit, patients who have not completed the screening will be randomized to receive a reminder to complete the mt-sDNA screening by one of three mechanisms (time 0):

1. Automated reminder using the EHR patient portal messaging system.
2. Automated reminder using a customized interactive voice response (IVR) system
3. Personalized reminder phone calls from the clinical team

This will allow for an empirical test of processes that can be employed to improve delivery of CRC screening and reduce preventable deaths in populations that are underserved with evidence-based interventions.

ELIGIBILITY:
Inclusion Criteria:

* Adults, between 50 to 75 years old.
* Due for colorectal cancer screening based on not having a record of a colonoscopy within 10 years, sigmoidoscopy, or CT colonography within 5 years, mt-sDNA within 3 years, or FIT within 1 year.
* Asymptomatic for colorectal cancer such as rectal bleeding or reported abdominal mass.

Exclusion Criteria:

* For the intervention study, patients will be restricted to those aged 50 to 75 years and are due for colorectal cancer screening.
* We will exclude any patient who has:
* Had prior colonoscopy within 10 years, sigmoidoscopy within 5 years, mt-sDNA within 3 years, CT colonography within 5 years, and FOBT/FIT within twelve months of inclusion into the study;
* A diagnosis of CRC or other GI cancer;
* History of confirmed Inflammatory Bowel Disease (Crohn's disease, ulcerative colitis) or other colitis;
* Had a colectomy, partial or total;
* A diagnosis of Lynch Syndrome;
* A diagnosis of Familial Adenomatous Polyposis (FAP);
* Iron deficiency anemia;
* Lower GI bleeding;
* A metastatic (Stage IV) blood or solid tumor cancer;
* End stage renal disease;
* A first degree relative with CRC prior to age 50 or 2+ first degree relatives diagnosed at any age.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint (intention-to-treat) | Completion by 6 months post randomization
  The completion rate of mt-sDNA among eligible patients. The primary comparison will be the return rate compared across intervention arms.

SECONDARY OUTCOMES:
Secondary Outcome (per protocol analysis) | Completion by 6 months post randomization
  The completion rate of mt-sDNA among eligible patients. The comparison will be the return rate compared across intervention arms, excluding participants who received an alternative intervention due to not having appropriate portal access.

CONTACTS AND LOCATIONS:
Overall Officials: Chyke Doubeni, MBBS, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials